CLINICAL TRIAL: NCT03864744
Title: Hepatic Histology and Metabolism Following Total Pancreatectomy and
Brief Title: Hepatic Histology and Metabolism Following Total Pancreatectomy and Pancreaticoduodenectomy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other); University of Copenhagen (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-18010755
Record Dates: First submitted 2019-03-01; First posted 2019-03-06 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Total Pancreatectomy; Pancreaticoduodenectomy; Pancreatic Diabetes; Non-Alcoholic Fatty Liver Disease; Metabolic Complication; Diabetes Mellitus
Keywords: liver biopsy; Lipid metabolism; Glucose metabolism; Postoperative complications; Pancreatic surgery
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to investigate the development of NAFLD following total pancreatectomy and pancreaticoduodenectomy and to explore the histological and metabolic changes following the procedures.

DETAILED DESCRIPTION:
After total pancreatectomy patients are treated with exogenous insulin and pancreatic enzyme supplementation in order to treat the endocrine and exocrine insufficiencies inherently occurring postoperatively. In addition to secondary diabetes and insufficient digestive capacity, totally pancreatectomised patients face a high risk of developing non-alcoholic hepatic steatosis. Under normal circumstances non-alcoholic fatty liver disease is regarded as the hepatic manifestation of metabolic syndrome and pathophysiologically related to excess energy intake and insulin resistance resulting in fat accumulation in adipose tissue as well as in the liver. Thus, the high incidence of hepatic steatosis following total pancreatectomy is surprising as patients typically are lean, peripherally insulin sensitive and properly insulinised.Interestingly, the pancreatic hormone glucagon has been implicated in lipid metabolism and recent human data from studies investigating the effect of glucagon receptor antagonism suggest that glucagon signalling may be essential for maintaining a fat-free liver. This makes the investigators speculate that the decreased glucagon levels following pancreatic surgery may play a hitherto unrecognised role in the development of hepatic steatosis after the operation.

The study will include 33 patients scheduled for pancreatectomy (total or pancreaticoduodenectomy). They will be followed for one year. A liver biopsy will be collected during the operation on all patients. After 12 months, participants will undergo magnetic resonance spectroscopy and those who have hepatic lipid content ≥2% will undergo an ultrasound-guided percutaneous liver biopsy. Furthermore, all participants will undergo a metabolic evaulation after one year.

ELIGIBILITY:
Inclusion Criteria:

* Subject scheduled for total pancreatectomy or pancreaticoduodenectomy
* Informed consent signed prior to any study-related procedure

Exclusion Criteria:

* Known liver disease before total pancreatectomy or pancreaticoduodenectomy (excluding NAFLD)
* Severe co-morbid disease (besides from the indication for the pancreas surgery)
* Pregnancy
* Any condition that the investigator feels would interfere with the safety of the trial participation or the safety of the subject
* Metastatic disease

Percutaneous liver biopsy exclusion criteria (to be evaluated before last visit)

* MR spectroscopy demonstrating lipid content <2%
* Haemoglobin <6 mmol/L
* INR >1.5
* Trombocytes <40 × 109/L
* Skin infection in area where biopsy will be sampled

Ages: 18 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who undergo total pancreatectomy or pancreaticoduodenectomy at Rigshospitalet, Copenhagen.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in hepatic lipid content (steatosis) after total pancreatektomy or pancreaticoduodenectomy | Baseline and after 12 months.
  Evaluated by light microscopy of the liver biopsy

SECONDARY OUTCOMES:
Hepatic lipid content | After 12 months
  Evaluated by magnetic resonance spectroscopy
Diagnosis and grade of steatohepatitis (steatosis, ballooning and lobular inflammation) | Baseline and after 12 months.
  Evaluated by light microscopy of the liver biopsy
Fibrosis stage (Kleiner classification) | Baseline and after 12 months.
  Evaluated by light microscopy of the liver biopsy
NAFLD activity score (NAS) | Baseline and after 12 months.
  Evaluated by light microscopy of the liver biopsy
Liver steatosis | After 12 months.
  Measured by controlled attenuation parametre (Fibroscan) in decibel per meter (dB/m)
Liver stiffness | After 12 months
  Measured by transcient elastrography (Fibroscan) in kilopascals (kPa)
Pancreatic endocrine dysfunction | After 12 months
  defined by HbA1c ≥ 6.5% and/or need for diabetes therapy
Alpha- and beta cell function | After 12 months
  measured by arginine stimulation test
Pancreatic exocrine dysfunction | After 12 months
  defined by f-elastase < 100 μg/g
Blood markers of liver function | Baseline and after 12 months
  including alanine transaminase (ALAT), aspartate aminotransferase (ASAT), gamma-glutamyltransferase (GGT), alkaline phosphatase, lactate dehydrogenase and bilirubin
Blood markers of glucose metabolism | Baseline and after 12 months
  HbA1c
Blood markers of glucose metabolism | Baseline and after 12 months
  Insulin
Blood markers of glucose metabolism | Baseline and after 12 months
  C-peptide
Blood markers of glucose metabolism | Baseline and after 12 months
  Glucagon
Blood markers of lipid metabolism | Baseline and after 12 months
  including lipid profiling
Blood markers of protein metabolism | Baseline and after 12 months
  including fractionated amino acids
Blood markers of nutritional status | Baseline and after 12 months
  including vitamin E and D, trace elements, lymphocytes and albumin
Blood markers related to bile-acid metabolism | Baseline and after 12 months
  including complement 4 (C4) and fibroblast growth factor 19 (FGF-19)
Changes in NAFLD/NASH biomarkers | Baseline and after 12 months
  including FGF-21

CONTACTS AND LOCATIONS:
Overall Officials: Filip Krag Knop, Professor, Study Director — Steno Diabetes Center Copenhagen, Clinical metabolic physiology
Locations (1):
- Steno Diabetes Center Copenhagen, Hellerup, Denmark